CLINICAL TRIAL: NCT02612428
Title: A Randomized, Open-Label, Multicenter, Controlled, Pivotal Study to Assess Safety and Efficacy of ELAD in Subjects With Alcohol-Induced Liver Decompensation (AILD)
Brief Title: Randomized, Open-Label, Multicenter, Controlled, Pivotal Study to Assess Safety and Efficacy of ELAD in Subjects w/ AILD
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: VTL-308 failed to meet its primary endpoint, all follow up studies were terminated
Sponsor: Vital Therapies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VTL-308
Record Dates: First submitted 2015-11-19; First posted 2015-11-23 (Estimated); Results first posted 2019-01-25 (Actual); Last update posted 2019-01-25 (Actual); Status verified 2019-01

CONDITIONS: Acute Alcoholic Hepatitis
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ELAD System (Experimental): This group will receive treatment with ELAD plus standard of care therapy.
  Interventions: Biological: ELAD System
- Standard of Care (Control) (Other): This group will receive standard of care therapy as defined in the protocol.
  Interventions: Other: Standard of Care (Control)

INTERVENTIONS:
Biological: ELAD System — An extracorporeal human hepatic cell-based liver treatment
  Other Names: ELAD
  Arms: ELAD System
Other: Standard of Care (Control) — Standard medical treatment as defined by the protocol
  Other Names: Standard of Care
  Arms: Standard of Care (Control)

SUMMARY:
The primary objective of the study is to evaluate safety and efficacy of ELAD with respect to overall survival of subjects with a clinical diagnosis of alcohol-induced liver decompensation (AILD) through at least Study Day 91.

The secondary objective is to evaluate the proportion of survivors at Study Day 91 using a chi-squared test.

DETAILED DESCRIPTION:
The ITT population includes all randomized subjects assigned to the group to which they were randomized, irrespective of actual treatment administered. Participant, Baseline Characteristics, and Outcome Measures used the ITT population. The safety population is defined as all subjects who are randomized based on actual treatment received. All serious adverse events and all non-serious adverse events analyses used the safety population.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet ALL inclusion criteria to be eligible for the study:

1. Age ≥18;
2. Total bilirubin ≥16 mg/dL (≥273.6 µmol/L);
3. A clinical diagnosis of alcohol-induced liver decompensation (AILD), based upon lab test or medical history or family interview with a causal relationship and temporal association (6 weeks or less) of alcohol use and hospital admission for this episode of AILD;
4. Maddrey score ≥32;
5. Subjects must have AILD that is severe acute alcoholic hepatitis (sAAH) diagnosed with either:

   a. A confirmatory liver biopsy, OR b. Two or more of the following: i. Hepatomegaly, ii. AST > ALT, iii. Ascites, iv. Leukocytosis (WBC count above lab normal at site);

   Note: Subjects will be classified as either:
   1. AILD that is sAAH with no underlying liver disease other than alcoholic liver disease, OR
   2. AILD that is sAAH with evidence of underlying liver disease other than alcoholic liver disease which must be documented by:

   i. Liver biopsy, AND/OR ii. Laboratory findings, AND/OR iii. Medical history;
6. Not eligible for liver transplant during this hospitalization;
7. Subject or legally-authorized representative must provide Informed Consent;
8. Subject must be eligible for Standard of Care treatment as defined in the protocol.

Exclusion Criteria:

Subjects must NOT have any of the exclusion criteria to be eligible for the study:

1. Age ≥50;
2. Platelet count <40,000/mm3;
3. International Normalization Ratio (INR) >2.5;
4. Serum Creatinine ≥1.3 mg/dL (≥115.04 µmol/L);
5. MELD score ≥30;
6. AST >500 IU/L;
7. Evidence of infection unresponsive to antibiotics (e.g. increased tissue involvement relative to initial diagnosis, clinical worsening of symptoms, etc.) indicated by any of the following:

   1. Presence of sepsis or septic shock; OR
   2. Positive blood cultures (bacteremia, fungemia) within 72 hours prior to Randomization; OR
   3. Presence of spontaneous bacterial peritonitis during the 2 days prior to Randomization; OR
   4. Clinical and radiological signs of pneumonia;
8. Evidence of reduction in total bilirubin of 20% or more in the previous 72 hours. Bilirubin measurements must be taken at least 12 hours after any procedure known to artificially alter serum bilirubin (e.g., administration of packed red blood cells, plasma exchange);
9. Evidence of hemodynamic instability as defined by the following:

   1. Systolic blood pressure <90 mmHg with evidence of diminished perfusion unresponsive to fluid resuscitation and/or low-dose pressor support; OR
   2. Mean arterial pressure (MAP) <60 mmHg with evidence of diminished perfusion unresponsive to fluid resuscitation and/or low-dose pressor support; OR
   3. Requirement for escalating doses of vasopressor support prior to Screening; OR
   4. Subject on vasopressors, including but not limited to those listed below, at doses above the following at Screening or Randomization:

      * Dobutamine: 5.0 µg/kg/min
      * Dopamine: 2.0 µg/kg/min
      * Norepinephrine: 0.02 µg/kg/min
      * Phenylephrine: 1.0 µg/kg/min
      * Vasopressin: 0.02 U/min
10. Evidence of active bleeding, major hemorrhage defined as requiring ≥2 units packed red blood cells to maintain a stable hemoglobin occurring within 48 hours prior to Randomization, or with banding of gastroesophageal varices during the 7 days immediately preceding screening;
11. Clinical evidence of liver size reduction due to cirrhosis [liver size of the craniocaudal diameter (sagittal view) <10 cm when measured on the mid clavicular line (or equivalent measurement) by ultrasound, or liver volume <1200 cc as determined by CT or MRI], unless Investigator interpretation of the clinical evidence indicates liver size of <10 cm or volume <1200 cc is not considered reduced for the individual subject, and Sponsor agrees;
12. Occlusive portal vein thrombosis impairing hepatopetal flow, or evidence of bile duct obstruction;
13. Evidence by physical exam, history, or laboratory evaluation, of significant concomitant disease with a life expectancy of less than 3 months, including, but not limited to:

    1. Severe acute or chronic cardiovascular, central nervous system, or pulmonary disease;
    2. Cancer that has metastasized or has not yet been treated;
    3. Severe metabolic abnormalities that have not been corrected (See Section 5.1.3);
14. Subject has chronic end-stage renal disease requiring chronic hemodialysis for more than 8 weeks (not classified as hepatorenal syndrome);
15. Subject ventilated or intubated;
16. Subject on hemodialysis;
17. Subject has liver disease related to homozygous hemachromotosis, Wilson's disease, has non-alcoholic fatty liver disease, or Budd-Chiari Syndrome;
18. Serological evidence (including viral titers) of active viral hepatitis A, B or C infection. If the investigator suspects that the subject may be at risk for viral hepatitis A, B or C, and no serology is available, then serologies must be obtained prior to Randomization, as a positive serology would be exclusionary;
19. Pregnancy as determined by serum β-human chorionic gonadotropin (HCG) results, or subjects of child-bearing potential not willing to use effective means of contraception, without history of medical or surgical sterilization;
20. Participation in another investigational drug, biologic, or device study within one month of enrollment, except for observational studies (the observational study setting should not affect the safety and/or efficacy of the VTL-308 clinical trial);
21. Previous liver transplant;
22. Previous enrollment in the treatment phase of another ELAD trial;
23. Have a Do Not Resuscitate or a Do Not Intubate (DNR/DNI) directive (or such local equivalent) or any other Advanced Directive limiting Standard of Care in place (the DNR/DNI criterion is not applicable in Europe);
24. Refusal to participate in the VTL-308E follow-up study;
25. Inability to provide an address for home visits.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 151 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jan Stange, MD, Study Director — Vital Therapies, Inc.; David Reich, MD, Principal Investigator — PA - Drexel University; Lance Stein, MD, Principal Investigator — GA - Piedmont Atlanta Hospital; Nikolaos Pyrsopoulos, MD, Principal Investigator — NJ - Rutgers University Hospital; Valentin Cuervas-Mons, MD, Principal Investigator — Spain - Hospital Universitario Puerta de Hierro Majadahonda; Raza Malik, MD, Principal Investigator — MA - Beth Israel Deaconess Medical Center; Nikunj Shah, MD, Principal Investigator — IL - Rush University Medical Center; Simona Rossi, MD, Principal Investigator — PA - Albert Einstein Medical Center; Juan Caballeria, MD, Principal Investigator — Spain - Hospital Clinic de Barcelona; Ram Subramanian, MD, Principal Investigator — GA - Emory University Hospital; Andres Duarte-Rojo, MD, Principal Investigator — AR - University of Arkansas for Medical Sciences; Julie Thompson, MD, Principal Investigator — MN - University of Minnesota; Peter R Galle, MD, Principal Investigator — Germany - Universitätsmedizin Mainz; Hartmut H.-J. Schmidt, MD, Principal Investigator — Germany - Universitätsklinikum Münster; Markus Busch, MD, Principal Investigator — Germany - Medizinische Hochschule Hannover; Kristina Chacko, MD, Principal Investigator — NY - Montefiore Medical Center; Talal Adhami, MD, Principal Investigator — OH - Cleveland Clinic Foundation; Constance Mobley, MD, PhD, Principal Investigator — TX - Houston Methodist Hospital; David J Kramer, MD, Principal Investigator — WI - Aurora St. Luke's Medical Center; Stephen Caldwell, MD, Principal Investigator — VA - University of Virginia Health System; Ali Al-Khafaji, MD, Principal Investigator — PA - University of Pittsburgh Medical Center; Kalyan R Bhamidimarri, MD, Principal Investigator — FL - Schiff Center for Liver Diseases/University of Miami; Manuel Romero-Gomez, MD, Principal Investigator — Spain - Hospital Universitario Virgen del Rocío; Tarek Hassanein, MD, Principal Investigator — CA - Sharp Coronado Hospital; Waldo Concepcion, MD, Principal Investigator — CA - Stanford University Medical Center; Martin Prieto Castillo, MD, Principal Investigator — Spain - Hospital Universitario y Politécnico La Fe; Rafael Bañares, MD, Principal Investigator — Spain - Hospital Universitario Gregorio Marañón; Syed Naqvi, MD, Principal Investigator — MO - University of Missouri Hospital; Matthias Dollinger, MD, PhD, Principal Investigator — Germany - Klinikum Landshut gemeinnuetzige GmbH; Karen Krok, MD, Principal Investigator — PA - The Pennsylvania State University and The Milton S. Hershey Medical Center; Rudolf Stauber, MD, Principal Investigator — Austria - Medizinische Universität Graz; Christian Zauner, MD, Principal Investigator — Austria - Medizinische Universität Klinik Für Innere Medizin III; Georg Lamprecht, MD, Principal Investigator — Germany - Universitätsmedizin Rostock; Paul Thuluvath, MD, Principal Investigator — MD - Mercy Medical Center; Trinidad Serrano Aullo, MD, Principal Investigator — Spain - Hospital Clínico Universitario Lozano Blesa
Locations (44):
- United States (21):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Sharp Coronado Hospital, Coronado, California
  - Stanford University Medical Center, Palo Alto, California
  - Schiff Center for Liver Diseases/University of Miami, Miami, Florida
  - Piedmont Atlanta Hospital, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Mercy Medical Center, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - University of Missouri Hospital, Columbia, Missouri
  - Rutgers University Hospital, Newark, New Jersey
  - Montefiore Medical Center, The Bronx, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - The Pennsylvania State University and The Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Drexel University, Philadelphia, Pennsylvania
  - Albert Einstein Medical Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Houston Methodist Hospital, Houston, Texas
  - University of Virginia Health System, Charlottesville, Virginia
  - Aurora St. Luke's Medical Center, Milwaukee, Wisconsin
- Austria (2):
  - Medizinische Universität Graz, Graz, Styria
  - Medizinische Universität Klinik Für Innere Medizin III, Vienna
- Germany (5):
  - Klinikum Landshut gemeinnuetzige GmbH, Landshut, Bavaria
  - Medizinische Hochschule Hannover, Hanover
  - Universitätsmedizin Mainz, Mainz
  - Universitätsklinikum Münster, Münster
  - Universitätsmedizin Rostock, Rostock
- St. Vincent's University Hospital, Dublin, Ireland
- Spain (6):
  - Hospital Puerta de Hierro Majadahonda, Majadahonda, Madrid
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitario Gregorio Marañón, Madrid
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Universitario y Politécnico La Fe, Valencia
  - Hospital Clínico Universitario Lozano Blesa, Zaragoza
- United Kingdom (9):
  - Aintree University Hospital, Liverpool, England
  - Ninewells Hospital and Medical School, Dundee, Scotland
  - Glasgow Royal Infirmary, Glasgow, Scotland
  - Belfast Health and Social Care Trust, Belfast
  - Queen Elizabeth Hospital, Birmingham
  - Doncaster Royal Infirmary, Doncaster
  - Royal London Hospital, London
  - Royal Free Hospital, London
  - Nottingham University Hospital, Nottingham

REFERENCES:
- See also: Company website — http://vitaltherapies.com

RESULTS

PARTICIPANT FLOW:
Period: VTL-308
Arm/Group | ELAD System | Standard of Care (Control)
Started | 78 | 73
Completed | 64 | 56
Not Completed | 14 | 17
Not completed — Death | 14 | 16
Not completed — Withdrawal by Subject | 0 | 1
Period: VTL-308E
Arm/Group | ELAD System | Standard of Care (Control)
Started | 64 | 56
Completed | 53 | 49
Not Completed | 11 | 7
Not completed — Death | 9 | 7
Not completed — Lost to Follow-up | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ELAD System | Standard of Care (Control) | Total
Number analyzed (Participants) | 78 | 73 | 151
Age, Customized [Count of Participants; unit: Participants]
  Age: Between 18 and 35 years | 23 | 22 | 45
  Age: Between 36 and 50 years | 55 | 51 | 106
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 29 | 60
  Male | 47 | 44 | 91
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 2 | 7
  White | 70 | 67 | 137
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  Austria | 0 | 2 | 2
  United States | 57 | 52 | 109
  Ireland | 1 | 0 | 1
  United Kingdom | 11 | 11 | 22
  Germany | 4 | 5 | 9
  Spain | 5 | 3 | 8
Baseline MELD Score [Mean (Standard Deviation); unit: MELD Score] — Measure Description: A higher baseline Model for End-stage Liver Disease (MELD) score value represents a worse outcome. The full theoretical scale range for MELD scores is from 6 to 40. This study excluded subjects with MELD score ≥30 according to the Protocol. In this study, the Min/Max MELD score in all subjects was 19/29.
  MELD Score | 24.8 (2.37) | 25.6 (2.35) | 25.2 (2.38)

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: The primary endpoint of the study was a comparison of overall survival (OS) between the ELAD-treated and Control groups, with protocol VTL-308E providing additional survival data up to a maximum of 5 years, that was included as available at the time of database lock (28 Aug 2018).
Time Frame: Up to at least Study Day 91, with protocol VTL-308E providing additional survival data (at 6, 9, 12, 24 months) at the time of database lock (28 August 2018).
Measure: Count of Participants; unit: Participants
Arm/Group | ELAD System | Standard of Care (Control)
Number analyzed (Participants) | 78 | 73
Participants | 55 | 51
Statistical Analysis 1: Comparison: ELAD System vs Standard of Care (Control); The primary endpoint was assessed using a Kaplan-Meier survival analysis of the Intent-to-treat (ITT) population utilizing a log-rank test; Test type: Superiority; p = 0.762, Log Rank; Hazard Ratio (HR) = 0.913, 95% CI 2-sided [0.509 to 1.640]

2. Secondary Outcome: Number of Survivors at Study Day 91
Description: Assess the proportion of survivors at Study Day 91
Time Frame: Up to Study Day 91
Measure: Count of Participants; unit: Participants
Arm/Group | ELAD System | Standard of Care (Control)
Number analyzed (Participants) | 78 | 73
Participants | 63 | 57
Statistical Analysis 1: Comparison: ELAD System vs Standard of Care (Control); Test type: Superiority; p = 0.6829, Chi-squared

3. Secondary Outcome: Number of Subjects With Early Change in Bilirubin Levels at Study Day 7
Description: To estimate the effect of ELAD on the number of subjects achieving a 20% reduction in total bilirubin by Day 7 (ECBL20 Yes)
Time Frame: Up to Study Day 7
Measure: Count of Participants; unit: Participants
Arm/Group | ELAD System | Standard of Care (Control)
Number analyzed (Participants) | 78 | 73
Participants | 38 | 24
Statistical Analysis 1: Comparison: ELAD System vs Standard of Care (Control); Test type: Superiority; p = 0.048, Chi-squared

ADVERSE EVENTS:
Time Frame: Randomization through Study Day 91.
Description: According to the SAP, Safety Population was used for the analysis of all adverse events and the Safety Population was defined according to the actual treatment received. Two subjects were not treated with ELAD because they did not meet the safety eligibility criteria before the start of ELAD treatment and they were included in the Control group in the Safety Population. Therefore, only 76 subjects were exposed to ELAD treatment and 75 subjects were exposed to Control.
Arm/Group | ELAD System | Standard of Care (Control)
All-Cause Mortality (participants affected / at risk) | 14/76 | 17/75
Serious Adverse Events (participants affected / at risk) | 47/76 | 42/75
Other Adverse Events (participants affected / at risk) | 76/76 | 74/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ELAD System (N=76) | Standard of Care (Control) (N=75)
Anaemia (Blood and lymphatic system disorders) | 4 (5) | 3 (4)
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Pulseless Electrical Activity (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 2 (2) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 3 (4) | 1 (1)
Alcoholic Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 4 (4)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 6 (7) | 7 (7)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Peritoneocutaneous Fistule (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Generalised Oedema (General disorders) | 1 (1) | 1 (1)
Medical Device Site Haematoma (General disorders) | 1 (1) | 0 (0)
Medical Device Haemorrhage (General disorders) | 1 (1) | 0 (0)
Multi-Organ Failure (General disorders) | 7 (7) | 13 (13)
Oedema Peripheral (General disorders) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Systemic Inflammatory Response Syndrome (General disorders) | 2 (2) | 1 (1)
Alcoholic Liver Disease (Hepatobiliary disorders) | 1 (1) | 1 (1)
Bioduct Stone (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic Cirrhosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic Failure (Hepatobiliary disorders) | 6 (6) | 5 (5)
Hepatic Function Abnormal (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatitis Alcoholic (Hepatobiliary disorders) | 3 (3) | 4 (4)
Hepatorenal Failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatorenal Syndrome (Hepatobiliary disorders) | 7 (7) | 5 (5)
Anaphylactoid Reaction (Immune system disorders) | 2 (2) | 0 (0)
Drug Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 3 (3) | 3 (3)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0)
Peritonitis Bacterial (Infections and infestations) | 0 (0) | 2 (2)
Pneumonia (Infections and infestations) | 4 (5) | 5 (6)
Sepsis (Infections and infestations) | 1 (1) | 1 (1)
Sepsis Syndrome (Infections and infestations) | 1 (1) | 0 (0)
Septic Shock (Infections and infestations) | 4 (4) | 4 (4)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 1 (1)
Head Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post-Procedural Haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Metabolic Acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Demyelination (Nervous system disorders) | 0 (0) | 1 (1)
Hepatic Encephalopathy (Nervous system disorders) | 2 (3) | 7 (8)
Seizure (Nervous system disorders) | 1 (1) | 1 (1)
Subarachnoid Haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Adjustment Disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Alcohol Abuse (Psychiatric disorders) | 1 (1) | 1 (1)
Alcohol Withdrawal Syndrome (Psychiatric disorders) | 2 (2) | 0 (0)
Acute Kidney Injury (Renal and urinary disorders) | 7 (8) | 6 (7)
Renal Failure (Renal and urinary disorders) | 2 (2) | 1 (1)
Renal Tubular Necrosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary Retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal Haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Hepatic Hyrdothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Respiratory Arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oesophageal Variceal Ligation (Surgical and medical procedures) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 3 (3)
Hypovolaemic Shock (Vascular disorders) | 1 (1) | 2 (2)
Orthostatic Hypotenstion (Vascular disorders) | 0 (0) | 1 (1)
Shock (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ELAD System (N=76) | Standard of Care (Control) (N=75)
Abdominal Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acquired Disfibrinogenaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 37 (42) | 18 (19)
Coagulopathy (Blood and lymphatic system disorders) | 14 (15) | 10 (10)
Disseminated Intravascular Coagulation (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Hypofibrinogenaemia (Blood and lymphatic system disorders) | 5 (6) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 13 (13) | 15 (16)
Lymphademopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Neutrophelia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 17 (18) | 8 (8)
Aortic Valve Incompetence (Cardiac disorders) | 0 (0) | 1 (1)
Atrial Fibrilation (Cardiac disorders) | 1 (1) | 1 (1)
Atrial Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 2 (2) | 2 (2)
Cardiac Failure Congestive (Cardiac disorders) | 2 (2) | 0 (0)
Cardiomegaly (Cardiac disorders) | 1 (1) | 0 (0)
Cardiovascular Disorder (Cardiac disorders) | 0 (0) | 1 (1)
Defect Conduction Intraventricular (Cardiac disorders) | 0 (0) | 1 (1)
Dilatation Ventricular (Cardiac disorders) | 1 (1) | 0 (0)
Heart Valve Incompetence (Cardiac disorders) | 2 (2) | 0 (0)
Left Atrial Dilatation (Cardiac disorders) | 2 (2) | 1 (1)
Left Ventricular Dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial Infarction (Cardiac disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Right Atrial Dilatation (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 9 (9) | 8 (8)
Tricuspid Valve Incompetence (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular Extrasystoles (Cardiac disorders) | 0 (0) | 2 (2)
Middle Ear Effusion (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Adrenal Insufficiency (Endocrine disorders) | 1 (1) | 2 (2)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Secondary Adrenocortical Insufficiency (Endocrine disorders) | 0 (0) | 1 (1)
Dry Eye (Eye disorders) | 3 (3) | 0 (0)
Vision Blurred (Eye disorders) | 1 (1) | 0 (0)
Vitreous Floaters (Eye disorders) | 0 (0) | 1 (1)
Abdominal Distension (Gastrointestinal disorders) | 2 (2) | 3 (3)
Abdominal Pain (Gastrointestinal disorders) | 16 (21) | 15 (18)
Anal Fissure (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anorectal Discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anorectal Varices (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 14 (14) | 22 (22)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 5 (5) | 6 (7)
Diarrhoea (Gastrointestinal disorders) | 26 (29) | 19 (19)
Diverticulum (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dry Mouth (Gastrointestinal disorders) | 3 (3) | 0 (0)
Duodenal Ulcer (Gastrointestinal disorders) | 2 (2) | 1 (1)
Duodenitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 3 (3)
Fecal Incontinence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastric Entral Vascular Ectasia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric Haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric Mucosal Lesion (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric Ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric Varices (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 3 (3)
Gastritis Erosive (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 11 (12) | 10 (10)
Gastrointestinal Mucosa Hyperaemia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 4 (4) | 0 (0)
Gingival Pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 3 (3)
Haemorrhoids (Gastrointestinal disorders) | 6 (6) | 2 (2)
Hiatus Hernia (Gastrointestinal disorders) | 2 (2) | 2 (2)
Ileus (Gastrointestinal disorders) | 2 (2) | 2 (2)
Ileus Paralytic (Gastrointestinal disorders) | 2 (2) | 0 (0)
Inguinal Hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large Intestine Polyp (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lip Dry (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mesenteric Haematoma (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 19 (20) | 13 (14)
Oesophageal Ulcer (Gastrointestinal disorders) | 2 (2) | 2 (2)
Oesophagitis (Gastrointestinal disorders) | 2 (2) | 1 (1)
Oesophagitis Ulcerative (Gastrointestinal disorders) | 0 (0) | 1 (1)
Painful Defaecation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Pacreatolithiasis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Periodontal Disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Peritoneal Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Peritonealcutaneous Fistula (Gastrointestinal disorders) | 1 (1) | 1 (1)
Portal Hypertensive Gastropathy (Gastrointestinal disorders) | 8 (8) | 8 (8)
Proctalgia (Gastrointestinal disorders) | 1 (1) | 1 (2)
Rectal Fissure (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal Haemorrhage (Gastrointestinal disorders) | 2 (2) | 1 (1)
Retroperitoneal Haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 2 (2) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0)
Umbilical Hernia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Varices Oesophageal (Gastrointestinal disorders) | 7 (7) | 9 (11)
Vomiting (Gastrointestinal disorders) | 16 (17) | 7 (10)
Abasia (General disorders) | 0 (0) | 1 (1)
Adverse Drug Reaction (General disorders) | 1 (1) | 1 (1)
Application Site Dysaesthesia (General disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 2 (3) | 1 (1)
Catheter Site Haemorrhage (General disorders) | 4 (4) | 3 (5)
Catheter Site Pain (General disorders) | 3 (4) | 4 (4)
Catheter Site Pruritus (General disorders) | 1 (1) | 0 (0)
Chest Pain (General disorders) | 1 (1) | 1 (1)
Chills (General disorders) | 2 (2) | 2 (2)
Fatigue (General disorders) | 3 (3) | 4 (4)
Gait Disturbance (General disorders) | 1 (2) | 1 (1)
Generalised Oedema (General disorders) | 6 (6) | 7 (7)
Hypothermia (General disorders) | 1 (1) | 2 (2)
Localised Oedema (General disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 1 (1) | 0 (0)
Medical Device Complication (General disorders) | 1 (1) | 0 (0)
Medical Device Site Haemorrhage (General disorders) | 14 (15) | 0 (0)
Medical Device Site Pain (General disorders) | 11 (11) | 0 (0)
Mucosal Inflammation (General disorders) | 1 (1) | 0 (0)
Multi-Organ Failure (General disorders) | 0 (0) | 1 (1)
Non-Cardiac Chest Pain (General disorders) | 2 (2) | 0 (0)
Oedema (General disorders) | 4 (4) | 1 (1)
Oedema Peripheral (General disorders) | 20 (24) | 14 (19)
Pain (General disorders) | 5 (5) | 2 (3)
Pneumatosis (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 19 (21) | 16 (17)
Systemic Inflammatory Response Syndrome (General disorders) | 1 (1) | 2 (2)
Temperature Intolerance (General disorders) | 1 (1) | 0 (0)
Thrombosis in Device (General disorders) | 2 (2) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 2 (2) | 0 (0)
Cholestasis (Hepatobiliary disorders) | 1 (1) | 2 (2)
Gall Bladder Polyp (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic Cirrhosis (Hepatobiliary disorders) | 2 (2) | 2 (2)
Hepatorenal Syndrome (Hepatobiliary disorders) | 3 (3) | 6 (6)
Hypertransaminasaemia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Jaundice (Hepatobiliary disorders) | 2 (2) | 0 (0)
Portal Hypertension (Hepatobiliary disorders) | 3 (3) | 0 (0)
Portal Vein Thrombosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Anaphylactic Reaction (Immune system disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 1 (1)
Bacteraemia (Infections and infestations) | 11 (11) | 8 (8)
Bacterial Vaginosis (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (2) | 2 (2)
Candida Infection (Infections and infestations) | 4 (4) | 1 (1)
Catheter Site Infection (Infections and infestations) | 0 (0) | 2 (2)
Cellulitis (Infections and infestations) | 2 (3) | 2 (2)
Clostridium Difficile Colitis (Infections and infestations) | 2 (2) | 4 (4)
Cystitis (Infections and infestations) | 0 (0) | 1 (1)
Cytomegalovirus Viraemia (Infections and infestations) | 1 (1) | 0 (0)
Device Related Infection (Infections and infestations) | 2 (2) | 0 (0)
Device Related Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Endocarditis (Infections and infestations) | 0 (0) | 1 (1)
Enterococcal Infection (Infections and infestations) | 2 (2) | 0 (0)
Fungal Skin Infection (Infections and infestations) | 1 (1) | 0 (0)
H1N1 Influenza (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 1 (1)
Lower Respiratory Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Oesophageal Candidiasis (Infections and infestations) | 0 (0) | 2 (2)
Oral Candidiasis (Infections and infestations) | 2 (2) | 2 (2)
Oral Herpes (Infections and infestations) | 0 (0) | 1 (1)
Oropharyngeal Candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 0 (0) | 1 (1)
Peritonitis Bacterial (Infections and infestations) | 6 (6) | 4 (4)
Pneumonia (Infections and infestations) | 8 (8) | 7 (8)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Pyuria (Infections and infestations) | 1 (1) | 0 (0)
Respiratory Tract Infection Viral (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 4 (4) | 4 (4)
Septic Shock (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 2 (2) | 1 (1)
Tinea Cruris (Infections and infestations) | 0 (0) | 1 (1)
Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary Tract Infection (Immune system disorders) | 14 (15) | 10 (11)
Anal Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 7 (8) | 2 (2)
Corrosive Gastritis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Craniocerebral Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Endotracheal Intubation Complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Excoriation (Injury, poisoning and procedural complications) | 6 (6) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 4 (6) | 1 (1)
Head Injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Joint Injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Limb Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lip Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Muscle Strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post Procedural Discomfort (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Procedural Complication (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Procedural Pain (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Scratch (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Scrotal Haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin Abrasion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Skin Wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Suture Related Complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tooth Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Transfusion Reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
VIIth Nerve Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular Pseudoaneurysm (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine Aminotransferase Increased (Investigations) | 0 (0) | 1 (1)
Aspartate Aminotransferase Increased (Investigations) | 2 (2) | 0 (0)
Blood Lactate Dehydrogenase Increased (Investigations) | 3 (3) | 0 (0)
Blood Magnesium Decreased (Investigations) | 0 (0) | 1 (1)
Blood Pressure Decreasd (Investigations) | 1 (1) | 0 (0)
Breath Sounds Abnormal (Investigations) | 1 (2) | 2 (2)
Cardiac Murmur (Investigations) | 3 (3) | 6 (6)
Electrocardiogram QT Prolonged (Investigations) | 2 (2) | 1 (1)
Influenza B Virus Test Positive (Investigations) | 0 (0) | 1 (1)
Intra-Abdominal Pressure Increased (Investigations) | 1 (1) | 0 (0)
Ultrasound Abdomen Abnormal (Investigations) | 1 (1) | 0 (0)
Weight Decreased (Investigations) | 0 (0) | 1 (1)
Weight Increased (Investigations) | 1 (1) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Decreased Appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 4 (4) | 2 (2)
Diabetes Mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Fluid Overload (Metabolism and nutrition disorders) | 4 (4) | 5 (5)
Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperammonaemia (Metabolism and nutrition disorders) | 5 (5) | 6 (6)
Hypercalcaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 13 (15) | 7 (7)
Hyperkalaemia (Metabolism and nutrition disorders) | 9 (9) | 5 (5)
Hypermagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyernatraemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hyperphosphataemia (Metabolism and nutrition disorders) | 2 (2) | 4 (4)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 (3) | 3 (4)
Hypocalcaemia (Metabolism and nutrition disorders) | 4 (4) | 2 (2)
Hypoglycaemia (Metabolism and nutrition disorders) | 4 (5) | 4 (4)
Hypokalaemia (Metabolism and nutrition disorders) | 9 (11) | 12 (12)
Hypomagnesaemia (Metabolism and nutrition disorders) | 12 (12) | 8 (8)
Hyponatraemia (Metabolism and nutrition disorders) | 10 (11) | 6 (7)
Hypophosphataemia (Metabolism and nutrition disorders) | 18 (21) | 11 (11)
Hypovolaemia (Metabolism and nutrition disorders) | 4 (4) | 2 (2)
Lactic Acidosis (Metabolism and nutrition disorders) | 4 (4) | 5 (5)
Malnutrition (Metabolism and nutrition disorders) | 2 (2) | 3 (3)
Metabolic Acidosis (Metabolism and nutrition disorders) | 10 (12) | 3 (4)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Refeeding Syndrome (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Type 2 Diabetes Mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Vitamin A Deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Vitamin D Deficiency (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Athralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Back Pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 4 (4)
Exostosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Flank Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint Stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint Swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 7 (8) | 3 (3)
Sarcopenia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Asterixis (Nervous system disorders) | 2 (2) | 1 (1)
Central Nervous System Lesion (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral Atrophy (Nervous system disorders) | 1 (1) | 0 (0)
Disturbance in Attention (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 8 (8) | 3 (3)
Dysarthria (Nervous system disorders) | 0 (0) | 1 (1)
Generalised Tonic-Colonic Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 9 (10) | 2 (2)
Hemiparesis (Nervous system disorders) | 1 (1) | 0 (0)
Hepatic Encephalopathy (Nervous system disorders) | 27 (28) | 22 (25)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1)
Loss of Consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Metabolic Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Neuropathy Peripheral (Nervous system disorders) | 0 (0) | 1 (1)
Nystagmus (Nervous system disorders) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Peroneal Nerve Palsy (Nervous system disorders) | 1 (1) | 0 (0)
Polyneuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Quadriparesis (Nervous system disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 2 (3) | 2 (2)
Speech Disorder (Nervous system disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 4 (4) | 1 (1)
Abnormal Dreams (Psychiatric disorders) | 0 (0) | 1 (1)
Acute Stress Disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Adjustment Disorder with Depressed Mood (Psychiatric disorders) | 2 (2) | 0 (0)
Agitation (Psychiatric disorders) | 7 (7) | 7 (7)
Alcohol Withdrawal Syndrome (Psychiatric disorders) | 3 (3) | 0 (0)
Anxiety (Psychiatric disorders) | 8 (8) | 4 (4)
Confusional State (Psychiatric disorders) | 1 (1) | 2 (2)
Delirium (Psychiatric disorders) | 2 (2) | 1 (1)
Depressed Mood (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 3 (3) | 2 (2)
Disorientation (Psychiatric disorders) | 2 (2) | 0 (0)
Hallucination (Psychiatric disorders) | 0 (0) | 1 (1)
Hallucination, Visual (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 13 (13) | 9 (9)
Nervousness (Psychiatric disorders) | 1 (1) | 0 (0)
Panic Attack (Psychiatric disorders) | 2 (2) | 1 (1)
Sleep Disorder (Psychiatric disorders) | 1 (1) | 2 (2)
Acute Kidney Injury (Renal and urinary disorders) | 13 (14) | 17 (21)
Anuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Chromaturia (Renal and urinary disorders) | 2 (2) | 0 (0)
Dysuria (Renal and urinary disorders) | 2 (2) | 0 (0)
Nephropathy Toxic (Renal and urinary disorders) | 0 (0) | 1 (1)
Oliguria (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal Failure (Renal and urinary disorders) | 7 (7) | 4 (4)
Renal Impairement (Renal and urinary disorders) | 2 (2) | 1 (1)
Renal Salt-Wasting Syndrome (Renal and urinary disorders) | 0 (0) | 1 (1)
Urethro Prolapse (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary Incontinence (Renal and urinary disorders) | 0 (0) | 5 (5)
Urinary Retention (Renal and urinary disorders) | 0 (0) | 3 (3)
Amenorrhoea (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Erectile Dysfunction (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Genital Rash (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Gynecomastia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Nipple Pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Scrotal Oedema (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Scrotal Pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vaginal Discharge (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vaginal Haemorrhage (Reproductive system and breast disorders) | 2 (2) | 1 (1)
Vulovaginal Pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Acquired Diaphragmatic Eventration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 10 (11) | 4 (4)
Bronchial Hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 10 (12) | 12 (12)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 16 (17) | 8 (8)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 5 (5)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Hepatic Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 14 (15) | 13 (15)
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 5 (5)
Lung Consolidation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lung Infiltration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal Dryness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Pharyngeal Erythema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3)
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary Mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 4 (4)
Rales (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (3)
Respiratory Acidosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sleep Apnoea Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (5)
Tracheal Fistula (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Upper Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 3 (4) | 7 (7)
Dermatitis Bullous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dry Skin (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1)
Acchymosis (Skin and subcutaneous tissue disorders) | 2 (3) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Facial Wasting (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Ingrowing Nail (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Leukoplakia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Palmar Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 16 (19) | 18 (18)
Rash (Skin and subcutaneous tissue disorders) | 6 (6) | 2 (2)
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Rash Morbilliform (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Rash Papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin Discolouration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin Irritation (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Spider Naevus (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Telangiectasia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Splenorenal Shunt (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Aortic Arteriosclerosis (Vascular disorders) | 0 (0) | 1 (1)
Deep Vein Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Distributive Shock (Vascular disorders) | 2 (2) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 2 (2)
Hypotension (Vascular disorders) | 21 (24) | 9 (10)
Hypovolaemic Shock (Vascular disorders) | 0 (0) | 2 (2)
Orthostatic Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Peripheral Artery Aneurysm (Vascular disorders) | 1 (1) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 1 (1)
Shock Haemorrhagic (Vascular disorders) | 0 (0) | 1 (1)
Thrombophlebitis Superficial (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2015-11-20): https://cdn.clinicaltrials.gov/large-docs/28/NCT02612428/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-24): https://cdn.clinicaltrials.gov/large-docs/28/NCT02612428/SAP_001.pdf